CLINICAL TRIAL: NCT04709796
Title: The Use of High Concentration Hyaluronic Acid (HA) Transfer Medium in Repeated Implantation Failure (RIF) Patients
Acronym: RIFLE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BC-08429
Record Dates: First submitted 2020-12-16; First posted 2021-01-14 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: IVF; Embryo Loss; Miscarriage, Recurrent
MeSH Terms: conditions — Embryo Loss; Abortion, Habitual

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group: EmbryoGlue (Experimental): Embryo transfer with EmbryoGlue®
  Interventions: Drug: EmbryoGlue®, Vitrolife
- Control group (Active Comparator): Conventional embryo transfer
  Interventions: Drug: Conventional Transfer

INTERVENTIONS:
Drug: EmbryoGlue®, Vitrolife — The intervention under study is the application of EmbryoGlue®, a class III medical device (CE Marked). EmbryoGlue® is a bicarbonate buffered medium containing recombinant human albumin, hyaluronan and gentamicin as an antibacterial agent.
  Arms: Intervention group: EmbryoGlue
Drug: Conventional Transfer — The control arm is the conventional embryo transfer without Embryo glue medium
  Arms: Control group

SUMMARY:
This is a pilot study with the aim to investigate the beneficial effect of bicarbonate buffered medium containing hyaluronan and recombinant human albumin (EmbryoGlue®, Vitrolife) in patients with documented repeated implantation failure on live birth per randomized subject as primary endpoint.

ELIGIBILITY:
Inclusion Criteria:

* The trial only includes women with a clinical indication for ART with a history of RIF defined as the absence of implantation after two consecutive cycles of IVF, ICSI or frozen embryo replacement cycles where the cumulative number of transferred embryos was no less than four for cleavage-stage embryos and no less than two for blastocysts, with all embryos being of good quality and of appropriate developmental stage.

Furthermore, other specific 'RIF' investigations were performed and treated if necessary:

* Normal hysteroscopy
* Normal karyotype of both parents
* Coagulation screening (Antitrombine II deficiency, Factor VIII augmentation, APC resistance, Factor V + Factor II augmentation, Protein S and C deficiency an homocysteine augmentation)
* Auto-immune screening (Lupus anticoagulant, Rheumatoid Factor, Anti-nuclear antibodies, Anti-cardiolipine antibodies and Glycoprotein-1-antibodies)

Exclusion Criteria:

* • Simultaneous participation in another clinical study

  * Untreated and uncontrolled thyroid dysfunction
  * Tumors of the ovary, breast, uterus, pituitary or hypothalamus
  * Abnormal (not menstrual) vaginal bleeding without a known/diagnosed cause
  * Ovarian cysts or enlarged ovaries
  * Malformations of the reproductive organs
  * Moderate or severe hepatic impairment
  * Current use of oral contraceptives, anti-psychotics, anti-epileptics or chemotherapy
  * Patients who undergo preimplantation genetic testing (PGT), fertility preservation or oocyte donation
  * Couples needing TESE/MESA material

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 178 (Estimated)
Dates: Start 2021-03-03 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Live birth | 9 months after embryo transfer
  live birth per randomized subject.

SECONDARY OUTCOMES:
positive hCG | 11 days (± 2 days) after embryo transfer.
  cumulative positive hCG rate confirmed by blood sample
ongoing pregnancy rate | between 6 and 8 weeks of gestation
  cumulative ongoing pregnancy rate per randomized subject, confirmed by ultrasound

CONTACTS AND LOCATIONS:
Overall Officials: Dominic Stoop, MD, Principal Investigator — University Hospital, Ghent
Locations (1):
- UZ Ghent, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: Undecided